CLINICAL TRIAL: NCT03439124
Title: A Multicentre, Randomized, Investigator-blind, Active-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Ceftobiprole Versus Intravenous Standard-of-care Cephalosporin Treatment With or Without Vancomycin in Pediatric Patients Aged From 3 Months to Less Than 18 Years With Hospital-acquired Pneumonia or Community-acquired Pneumonia Requiring Hospitalisation
Brief Title: Ceftobiprole in the Treatment of Pediatric Patients With Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPR-PIP-002
Record Dates: First submitted 2018-01-30; First posted 2018-02-20 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Community-acquired Pneumonia (CAP); Hospital-acquired Pneumonia (HAP)
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia | interventions — ceftobiprole medocaril; ceftobiprole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceftobiprole medocaril (Experimental): Ceftobiprole medocaril is the water-soluble prodrug of ceftobiprole, an advanced-generation cephalosporin developed for IV administration. Ceftobiprole is characterized by potent, broad-spectrum antimicrobial activity against both Gram-positive and Gram-negative pathogens.
  Interventions: Drug: ceftobiprole medocaril
- IV standard-of-care cephalosporin (Active Comparator): Ceftriaxone was used as standard-of-care cephalosporin for the treatment of CAP. It is a third-generation cephalosporin with activity against typical bacterial pathogens of CAP requiring hospitalization, and is widely used for the treatment of various bacterial infections in neonates, infants, children, and adults.
  Ceftazidime was used as standard-of-care cephalosporin for the treatment of HAP. It is also a third-generation cephalosporin, but with broader activity against Gram-negative aerobic bacilli, including Pseudomonas aeruginosa.
  Vancomycin is a glycopeptide antibiotic that is active against staphylococci, including methicillin-resistant Staphylococcus aureus (MRSA). At the discretion of the blinded investigator, patients received vancomycin in addition to the IV standard-of-care cephalosporin when MRSA was suspected or confirmed.
  Interventions: Drug: IV standard-of-care cephalosporin

INTERVENTIONS:
Drug: ceftobiprole medocaril — Ceftobiprole medocaril was administered at age-adjusted doses (10, 15 or 20 mg/kg) and infusion durations (2 or 4 hours) every 8 hours. The maximum dose, regardless of body weight, was 500 mg ceftobiprole every 8 hours (maximum total daily dose of 1500 mg ceftobiprole).
  After a minimum of 3 days of IV treatment, patients with sufficient improvement in disease signs and symptoms could be switched to an age-appropriate oral antibiotic to complete a total minimum of 7 days and a total maximum of 14 days' antibiotic treatment.
  Other Names: ceftobiprole
  Arms: Ceftobiprole medocaril
Drug: IV standard-of-care cephalosporin — Ceftriaxone was administered at 50 to 80 mg/kg IV as a single daily dose, up to a maximum dose of 2 g/day. The actual dose of ceftriaxone within this dose range was determined by the blinded investigator prior to first study drug administration and was not modified during subsequent study days.
  After a minimum of 3 days of IV treatment, patients with sufficient improvement in disease signs and symptoms could be switched to an age-appropriate oral antibiotic to complete a total minimum of 7 days and a total maximum of 14 days' antibiotic treatment.
  At the discretion of the blinded investigator, patients received vancomycin at a dose of 10 to 15 mg/kg IV every 6 hours, up to a maximum dose of 2 g/day, in addition to the IV standard-of-care cephalosporin when MRSA was suspected or confirmed.
  Arms: IV standard-of-care cephalosporin

SUMMARY:
This was a study of the safety and efficacy of ceftobiprole medocaril compared with intravenous (IV) standard-of-care cephalosporin treatment with or without vancomycin in pediatric patients with either hospital-acquired bacterial pneumonia (HAP) or community-acquired bacterial pneumonia (CAP) requiring hospitalization, and requiring intravenous (IV) antibiotic therapy.

DETAILED DESCRIPTION:
This was a randomized, investigator-blind, active-controlled multi-center study to evaluate the safety, tolerability, pharmacokinetics and efficacy of ceftobiprole medocaril compared with IV standard-of-care cephalosporin treatment with or without vancomycin in pediatric patients aged 3 months to less than 18 years with HAP or CAP requiring hospitalization and therapy with IV antibiotics. Randomization was stratified by four age groups (3 months to < 2 years; 2 years to < 6 years; 6 years to < 12 years; 12 years to < 18 years), and by diagnosis of HAP or CAP.

ELIGIBILITY:
Inclusion Criteria:

* Male of female aged 3 months to < 18 years with a body weight of at least 5 kg
* Diagnosis of either hospital-acquired pneumonia or community-acquired pneumonia requiring hospitalization and administration of IV antibiotic therapy
* New or progressive imaging findings consistent with bacterial pneumonia
* Requirement for IV antibacterial treatment for pneumonia
* Other inclusion criteria may apply

Exclusion Criteria:

* Known resistance of the causative pathogen to ceftobiprole or IV standard-of-care cephalosporin treatment (± vancomycin)
* On mechanical ventilation
* Chest trauma with severe lung contusion or flail chest
* Acute respiratory distress syndrome
* Empyema or lung abscess
* Anatomical bronchial obstruction
* Active or currently treated pulmonary tuberculosis
* Atypical bacterial pneumonia, or viral pneumonia without bacterial superinfection, or need for antibiotic coverage with a macrolide
* Pertussis, chemical pneumonitis, or cystic fibrosis
* Severe immunodeficiency
* Significant laboratory abnormalities including: Hematocrit <20%; absolute neutrophil count <0.5x10⁹/L; platelet count <50x10⁹/L; alanine aminotransferase, aspartate aminotransferase, or bilirubin >5 times the age-specific upper limit of normal;
* Creatinine clearance <50 mL/min/1.73 m²
* Use of systemic antimicrobial therapy for more than 24 hours in the 48 hours before randomization
* History of a previous clinically-relevant hypersensitivity or serious adverse reaction to beta lactam antibiotics or to vancomycin
* Poorly controlled seizure disorder
* Other exclusion criteria may apply

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, MD, Study Director — Basilea Pharmaceutica
Locations (19):
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv
  - Multiprofile Hospital for Active Treatment, Rousse
  - University Multiprofile Hospital for Active Treatment "Aleksandrovska", Sofia
- Georgia (6):
  - Amtel Hospital First Clinical LLC, Tbilisi
  - LTD High Technology Medical Center University Clinic, Tbilisi
  - JSC Evex Hospitals 1, Tbilisi
  - JSC Evex Hospitals 2, Tbilisi
  - Tbilisi State Medical University G. Zhvania Pediatric Academic Clinic, Tbilisi
  - Ltd Tbilisi Pediatric Private Clinic, Tbilisi
- Hungary (7):
  - Principal SMO Ltd., Baja
  - Semmelweis University, Budapest
  - Central Hospital of Southern Pest National Institute of Hematology and Infectious Diseases, Budapest
  - Bekes County Central Hospital, Gyula
  - Kanizsai Dorottya Hospital, Nagykanizsa
  - Fejer County St. Gyorgy University Teaching Hospital, Székesfehérvár
  - Torokbalint Pulmonology Institute, Törökbálint
- Romania (2):
  - Alessandrescu-Rusescu National Institute for Mother and Child Health, Bucharest
  - Sf. Maria" Children's Emergency Clinical Hospital, Iași

REFERENCES:
- [Derived] Rubino CM, Polak M, Schropf S, Munch HG, Smits A, Cossey V, Tomasik T, Kwinta P, Snariene R, Liubsys A, Gardovska D, Hornik CD, Bosheva M, Ruehle C, Litherland K, Hamed K. Pharmacokinetics and Safety of Ceftobiprole in Pediatric Patients. Pediatr Infect Dis J. 2021 Nov 1;40(11):997-1003. doi: 10.1097/INF.0000000000003296. PMID 34533489
- [Derived] Bosheva M, Gujabidze R, Karoly E, Nemeth A, Saulay M, Smart JI, Hamed KA. A Phase 3, Randomized, Investigator-blinded Trial Comparing Ceftobiprole With a Standard-of-care Cephalosporin, With or Without Vancomycin, for the Treatment of Pneumonia in Pediatric Patients. Pediatr Infect Dis J. 2021 Jun 1;40(6):e222-e229. doi: 10.1097/INF.0000000000003077. PMID 33480665

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 138 randomized patients received treatment
Groups:
- IV Standard-of-care Cephalosporin: Ceftriaxone was used as standard-of-care cephalosporin for the treatment of community-acquired pneumonia (CAP). It is a third-generation cephalosporin with activity against typical bacterial pathogens of CAP requiring hospitalization, and is widely used for the treatment of various bacterial infections in neonates, infants, children, and adults.
  Ceftazidime was used as standard-of-care cephalosporin for the treatment of hospital-acquired pneumonia (HAP). It is also a third-generation cephalosporin, but with broader activity against Gram-negative aerobic bacilli, including Pseudomonas aeruginosa.
  Vancomycin is a glycopeptide antibiotic that is active against staphylococci, including methicillin-resistant Staphylococcus aureus (MRSA). At the discretion of the blinded investigator, patients received vancomycin in addition to the IV standard-of-care cephalosporin when MRSA was suspected or confirmed.
Period: Overall Study
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin
Started | 94 | 44
Completed | 90 | 44
Not Completed | 4 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- IV Standard-of-care Cephalosporin: Ceftriaxone was used as standard-of-care cephalosporin for the treatment of CAP. It is a third-generation cephalosporin with activity against typical bacterial pathogens of CAP requiring hospitalization, and is widely used for the treatment of various bacterial infections in neonates, infants, children, and adults.
  Ceftazidime was used as standard-of-care cephalosporin for the treatment of HAP. It is also a third-generation cephalosporin, but with broader activity against Gram-negative aerobic bacilli, including Pseudomonas aeruginosa.
  Vancomycin is a glycopeptide antibiotic that is active against staphylococci, including MRSA. At the discretion of the blinded investigator, patients received vancomycin in addition to the IV standard-of-care cephalosporin when MRSA was suspected or confirmed.
- Total: Total of all reporting groups
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin | Total
Number analyzed (Participants) | 94 | 44 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 94 | 44 | 138
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.81 [0.6 to 17] | 6.95 [1 to 17] | 6.86 [0.6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 23 | 64
  Male | 53 | 21 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 94 | 43 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Infection type [Count of Participants; unit: Participants]
  Hospital-acquired pneumonia | 5 | 3 | 8
  Community-acquired pneumonia | 89 | 41 | 130

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Reported are adverse events (AEs) during the first 3 days of IV therapy and while patients were on IV therapy irrespective of when they switched to oral antibiotic treatment.
Time Frame: Analysis of AEs assessed during the first 3 days of IV therapy and while on IV, a median of 7 days
Population: Safety population: all randomized patients who received at least one dose of study drug, analyzed according to the first treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin
Number analyzed (Participants) | 94 | 44
Participants
  First 3 days of IV therapy: Non-Serious TEAE | 10 | 5
  First 3 days of IV therapy: Serious TEAE | 1 | 0
  First 3 days of IV therapy: TEAE leading to death | 0 | 0
  First 3 days of IV therapy: No TEAE | 83 | 39
  While on IV therapy: Non-Serious TEAE | 17 | 8
  While on IV therapy: Serious TEAE | 2 | 0
  While on IV therapy: TEAE leading to death | 0 | 0
  While on IV therapy: No TEAE | 75 | 36

2. Secondary Outcome: Proportion of Patients With Clinical Cure in the Intent-to-treat Population (ITT)
Description: Comparison of clinical cure rates (signs and symptoms of pneumonia normalized or improved such that no further antibiotic therapy was necessary, and stabilization or improvement of chest X-ray findings if these were available) in the ITT population between ceftobiprole and the comparator at the TOC visit.
Time Frame: At the test-of-cure (TOC) visit
Population: Intent-to-treat (ITT) population: all randomized patients, analyzed by treatment assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin
Number analyzed (Participants) | 94 | 44
Participants | 85 | 43

3. Secondary Outcome: Proportion of Patients With Clinical Cure in the Clinically Evaluable (CE) Population
Description: Comparison of clinical cure rates (signs and symptoms of pneumonia normalized or improved such that no further antibiotic therapy was necessary, and stabilization or improvement of chest X-ray findings if these were available) in the CE population between ceftobiprole and the comparator at the TOC visit.
Time Frame: At the TOC visit
Population: Clinically Evaluable (CE) population: all patients who had a valid clinical outcome assessment at TOC and no major protocol deviations such as non-study antibiotic therapies.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin
Number analyzed (Participants) | 88 | 41
Participants | 80 | 41

4. Secondary Outcome: Proportion of Patients With Early Clinical Response in the Intent-to-treat (ITT) Population
Description: Comparison of early clinical response rates in the ITT population between ceftobiprole and the comparator at Day 4.
Time Frame: At Day 4
Population: Intent-to-treat (ITT) population: all randomized patients, analyzed by treatment assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin
Number analyzed (Participants) | 94 | 44
Participants | 90 | 41

5. Secondary Outcome: Proportion of Patients With Early Clinical Response in the Clinically Evaluable (CE) Population
Description: Comparison of early clinical response rates in the CE population between ceftobiprole and the comparator at Day 4.
Time Frame: At Day 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin
Number analyzed (Participants) | 88 | 41
Participants | 84 | 39

ADVERSE EVENTS:
Time Frame: Relevant worsening of a patient's status after informed consent (before start of first study-drug infusion) was recorded in medical history. From start of first dosing to and including the last follow-up visit, 28 to 35 days after end-of-treatment, such worsening was recorded as an AE.
Description: Once an AE was detected, it was proactively followed up at each visit (or more frequently if necessary) for any changes in severity, relationship to the study drug, interventions required for treatment, and the event's outcome. Serious adverse events (SAEs) were to be additionally reported and recorded on SAE report forms.
Arm/Group | Ceftobiprole Medocaril | IV Standard-of-care Cephalosporin
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/44
Serious Adverse Events (participants affected / at risk) | 7/94 | 2/44
Other Adverse Events (participants affected / at risk) | 8/94 | 5/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftobiprole Medocaril (N=94) | IV Standard-of-care Cephalosporin (N=44)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftobiprole Medocaril (N=94) | IV Standard-of-care Cephalosporin (N=44)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT03439124/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03439124/SAP_001.pdf